CLINICAL TRIAL: NCT01889576
Title: The Effect of Magnesium Supplements on Early Post-transplantation Glucose Metabolism: a Randomized Controlled Trial.
Brief Title: The Effect of Magnesium on Early Post-transplantation Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDS BE-02-RG-219
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Glucose Metabolism After Transplantation
Keywords: glucose
MeSH Terms: interventions — Magnesium Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplementation of Magnesium oxide. (Experimental): Supplementation of magnesium oxide (450 mg up to 3 times daily maximum), aiming at a serum magnesium concentration of >= 1,9 mg/dL).
  Interventions: Dietary Supplement: Magnesium Oxide
- No supplementation or minimal dose. (No Intervention): No supplementation (or a minimal dose to keep serum magnesium concentration ≥ 1.2mg/dL depending on the treating physician).

INTERVENTIONS:
Dietary Supplement: Magnesium Oxide
  Arms: Supplementation of Magnesium oxide.

SUMMARY:
Hypomagnesemia is common early after transplantation, especially in association with calcineurin inhibitors and predicts diabetes after transplantation. Magnesium improves glycemic control and insulin sensitivity in diabetics and insulin resistant subjects without diabetes but this was never evaluated in transplant recipients.

The aim of the study is to assess whether magnesium improves glycemic control and insulin sensitivity early after transplantation.

The study is an open label study in which adult hypomagnesemic renal transplant recipients are randomized the first 2 weeks after kidney transplantation to magnesium oxide or no supplementation.

The hypothesis is that magnesium supplementation in renal transplant recipients exerts a beneficial effect on glycemia and the development of diabetes after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplantation recipients
* > 18 years of age
* Less than 2 weeks post-transplantation
* Hypomagnesemia < 1,7 milligram/deciliter on 2 consecutive blood samples (laboratory reference interval 1,7 - 2,55 milligram/deciliter).

Exclusion Criteria:

* Pre-existing diabetes mellitus defined as the intake of anti-diabetic drugs at the time of inclusion
* Serum creatinine > 3 milligram/deciliter
* Active infection (C reactive protein > 3 milligram/deciliter)
* Severe hypomagnesemia (< 1,2 milligram/deciliter)
* Hypokalemia (< 3,5 milli-equivalent/liter)
* Severe hypocalcemia (< 6,5 milligram/deciliter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fasting glycemia, 3 months after transplantation. | 3 months after transplantation.

SECONDARY OUTCOMES:
Incidence of diabetes after transplantation the first 3 months after transplantation. | 3 months after transplantation.
Incidence of impaired fasting glucose the first 3 months after transplantation. | 3 months after transplantation.
Insulin sensitivity measured by "Homeostatic Model assessment (HOMA)", 3 months after transplantation. | 3 months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Van Laecke, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Van Laecke S, Nagler EV, Taes Y, Van Biesen W, Peeters P, Vanholder R. The effect of magnesium supplements on early post-transplantation glucose metabolism: a randomized controlled trial. Transpl Int. 2014 Sep;27(9):895-902. doi: 10.1111/tri.12287. Epub 2014 Mar 24. PMID 24909487